CLINICAL TRIAL: NCT04415515
Title: Standard Care Coordination Expansion Pilot - A Quality Improvement Study
Brief Title: Standard Care Coordination Expansion Pilot
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Academic partnership between UHC and UCLA was terminated effective December 31, 2023
Sponsor: UnitedHealthcare (Other)
Collaborators: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Anthony Pirrello, Director UHC E&I Healthcare Econ, UnitedHealthcare
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: UHC100023A; DP006128 (Other Grant/Funding Number: CDC)
Record Dates: First submitted 2020-01-28; First posted 2020-06-04 (Actual); Last update posted 2025-11-12 (Actual); Status verified 2025-11

CONDITIONS: Superutilizers, Health Care Utilization
Keywords: Care coordination, case management, superutilizers, health care utilization
MeSH Terms: conditions — Patient Acceptance of Health Care | interventions — Disease Management

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Treatment 1 (Experimental): RN Standard care coordination and disease management + RN Case Management
  Interventions: Behavioral: RN case management; Behavioral: RN Standard care coordination and disease management
- Control (Experimental): RN Standard care coordination and disease management
  Interventions: Behavioral: RN Standard care coordination and disease management
- Treatment 2 (Experimental): RN Standard care coordination and disease management + Community Health Worker Case Management
  Interventions: Behavioral: Community Health Worker Case Management; Behavioral: RN Standard care coordination and disease management

INTERVENTIONS:
Behavioral: RN case management — A Registered Nurse (RN) case manager makes phone contact with the member to review medications, health risks, care gaps/barriers, & to develop a case management plan that focuses on improving medication adherence & reconciliation, condition-based measures & outcomes, addressing psycho-social needs, & intensive post-admission care transition. RNs may refer the member to social workers,specialist providers, & support programs (including to more intense case management where the primary care physician is notified that RNs may contact them to support treatment & coordinate services).
  Arms: Treatment 1
Behavioral: Community Health Worker Case Management — In selected UHC markets for defined time periods, members randomized to the treatment arm also received an enhanced version of the SCC that included in-home case management support from non-clinical Community Health Workers (CHW).
  Arms: Treatment 2
Behavioral: RN Standard care coordination and disease management — RN Standard care coordination and disease management

SUMMARY:
The Standard Care Coordination (SCC) solution integrates aspects of case management & care coordination & was designed by UnitedHealth Group for high-cost, complex, at-risk consumers to facilitate health care access and decisions that can have a dramatic impact on the quality and affordability of the consumer's health care. Currently members only receive the SCC if they are: 1) identified as high risk for readmission upon discharge from the hospital, 2) are self-referred, or 3) are directly referred to the program by their physician. The current quality improvement study was designed as a randomized controlled trial to determine if the expansion of the SCC program to commercially insured members identified via a proprietary administrative algorithms as being at high risk would significantly impact rates of acute inpatient admissions.

ELIGIBILITY:
Inclusion Criteria:

* UnitedHealthcare commercial Fully Insured members; all states; 18+ years old; actively enrolled in the health plan as of randomization identified via proprietary administrative algorithm as being at high risk for persistent super utilizer status.

Exclusion Criteria:

* : pregnant women, individuals prescribed medications for infertility, members with evidence of dementing disorders, members indicated as "do not contact " for program outreach, and Members in the following products and plans:

  * legacy UHC ASO groups (populations for which UHC provides administrative services only),
  * legacy Oxford health plan members (all members receive the SCC program),
  * legacy PacifiCare members,
  * legacy River Valley/NHP members, and
  * Public Sector clients
  * the PHS 2.0 intervention (a small population within Fully Insured)
  * assignment to a clinically activated Accountable Care Organization (ACO)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 592023 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2023-12 (Actual); Study Completion 2023-12 (Actual)

PRIMARY OUTCOMES:
Total Cost | 24 months
  Defined as total plan cost (medical and pharmacy) per member
Acute Inpatient Admission Rate | 24 months
  Defined as acute inpatient admissions per 1,000 qualified members
Emergency Room Visit Rate | 24 months
  Defined as the number of emergency room visits per 1,000 qualified members
Diabetes-Related Complications | 24 months
  Defined as the Diabetes Complications Severity Index (DCSI) composite score. The composite DCSI score ranges between 0 to 13 (sum of scores from 7 diabetes complication categories [cardiovascular disease, cerebrovascular disease/stroke, peripheral vascular disease, nephropathy, retinopathy, neuropathy, and metabolic complications such as ketoacidosis, hyperosmolar, or other coma] which are each scored from 0 to 2 [0=no complication, 1=non-severe complication, 2=severe complication], except for neuropathy which is scored from 0 to 1)

SECONDARY OUTCOMES:
Risk of Acute Inpatient Admission | 12, 18, 24, 36, 48 months
  Defined as time to first acute inpatient admission
All-Cause 30-Day Readmission Risk | 12, 18, 24, 36, 48 months
  Defined as first acute inpatient readmission for all-causes within 30 days of index acute inpatient discharge
Outpatient Emergency Room Visit Rate | 12, 18, 24, 36, 48 months
  Defined as emergency room visits per 1,000 qualified members per year
Risk of Emergency Room Visit | 12, 18, 24, 36, 48 months
  Defined as time to first emergency room visit
Primary Care Physician Visit Rate | 12, 18, 24, 36, 48 months
  Defined as primary care physician visits per qualified member
Specialist Physician Visit Rate | 12, 18, 24, 36, 48 months
  Defined as specialist physician visits per qualified member
Cardiovascular Disease | 12, 18, 24, 36, 48 months
  Defined as percentage of members with cardiovascular disease
Diabetes-related complications (DCSI) | 12, 18, 24, 36, 48 months
Amputations | 12, 18, 24, 36, 48 months
  Defined as lower extremity amputations per 1,000 qualified members
Chronic Kidney Disease | 12, 18, 24, 36, 48 months
  Defined as attenuated decline of eGFR, for members with baseline eGFR below 60mL/min
Glycemic Control | 12, 18, 24, 36, 48 months
  Defined as number of members with A1c below 7%, below 8%, and/or above 9%, per 100 qualified members with diabetes
Adherence to Diabetes-Related Medications | 12, 18, 24, 36, 48 months
  Defined as number of members with medication possession ratio (MPR) values of 80% or higher, per 100 qualified members with diabetes
Adherence to Diabetes-Related Processes of Care | 12, 18, 24, 36, 48 months
  Defined as rates of microalbuminuria screening, retinal/eye exams, A1c test frequency, LDL test frequency, Statin use, ACE/ARB use
Total Plan and Member Cost | 12, 18, 24, 36, 48 months
  Defined as total (plan+member) cost per member
Diabetes Complications Count | 12, 18, 24, 36, 48 months
  Defined as the Diabetes Complications Severity Index (DCSI) count. The DCSI count ranges from 0 to 7 (count of the 7 diabetes complication categories [cardiovascular disease, cerebrovascular disease/stroke, peripheral vascular disease, nephropathy, retinopathy, neuropathy, and metabolic complications such as ketoacidosis, hyperosmolar, or other coma]).
Any Acute Inpatient Admission | 12, 18, 24, 36, 48 months
  Defined as the number of members with any Acute Inpatient Admission per 1,000 qualified members
Any Emergency Room Visit | 12, 18, 24, 36, 48 months
  Defined as the number of members with any emergency room visit per 1,000 qualified members
Cerebrovascular disease/stroke | 12, 18, 24, 36, 48 months
  Defined as percentage of members with Cerebrovascular disease/stroke
Peripheral vascular disease | 12, 18, 24, 36, 48 months
  Defined as percentage of members with Peripheral vascular disease
Nephropathy | 12, 18, 24, 36, 48 months
  Defined as percentage of members with Nephropathy
Retinopathy | 12, 18, 24, 36, 48 months
  Defined as percentage of members with Retinopathy
Neuropathy | 12, 18, 24, 36, 48 months
  Defined as percentage of members with Neuropathy
Metabolic complications such as ketoacidosis, hyperosmolar, or other coma | 12, 18, 24, 36, 48 months
  Defined as percentage of members with metabolic complications

CONTACTS AND LOCATIONS:
Overall Officials: Anthony V Pirrello, MS, Principal Investigator — UnitedHealthcare
Locations (1):
- UnitedHealthcare, Minnetonka, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Duru OK, Harwood J, Moin T, Takada S, Tseng CH, Saju R, Lee E, Fatehpuria A, Mangione CM. Care Coordination for High-Need, High-Cost Commercially Insured Patients: A Randomized Clinical Trial. JAMA Netw Open. 2025 Jun 2;8(6):e2511804. doi: 10.1001/jamanetworkopen.2025.11804. PMID 40553475